CLINICAL TRIAL: NCT03285360
Title: Effectiveness of Sylc Air Abrasion Bioactive Glass Technology Versus Fluoride Varnish Application in Management of Hypersensitivity of Non-Carious Cervical Lesions: Randomized Clinical Trial.
Brief Title: Effectiveness of Bioactiveglass Air Abrasion Versus Fluoride Varnish in Management of Dentin Hypersensitivity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Ezz, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CairoU-DEzz
Record Dates: First submitted 2017-09-11; First posted 2017-09-18 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Hypersensitivity Dentin; Tooth Hypersensitivity
Keywords: Bifluoride, sylc, hypersensitivity,
MeSH Terms: conditions — Dentin Sensitivity; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Dentin Hypersensitivity
Who Masked: Participant, Outcomes Assessor
Masking Description: double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- sylc bioactive glass (Experimental): Sylc is a dry powder (calcium sodium phosphosilicate), based on NovaMin powder. Bottle of small and coarse particles will be used for the treatment.
  Steps:
  1. Isolation: D.M. will make proper isolation for the teeth using cotton rolls.
  2. Hand piece: NSK Prophymate Neo will be used to deliver the powder particles on the sensitive areas. Air stream adjusted at 40-46 psi.
  3. Application: The hand piece will be held at constant distance (3-4mm) away from the tooth surface, with 60-80 degrees on the buccal surfaces. The powder will be applied for 5-10 seconds per tooth in a circular movement.
  4. Suction: High volume suction will be used on lingual side of the teeth to suck any particles, and avoid patient from swallowing it.
  Interventions: Combination Product: Sylc
- fluoride varnish (Bifluorid 10) (Active Comparator): fluoride varnish Bifluorid 10(by VOCO) will be used. It is a rapid- drying suspension of equal amounts of sodium fluoride and calcium fluoride.
  The single dose form will be used, to make sure the amount of fluoride varnish used is standardized.
  Steps:
  1. Preparation: The tooth will be properly cleaned, and the surface will be air-dried.
  2. Dispensing: The foil will be pierced using a micro- tim, the opening will be enlarged, the brush will be wet in a circular movement.
  3. Application: Thin coat will be applied on the tooth surface. The varnish will be left from 10-20 seconds then air dried.
  Concerning the storage of the Bifluoride 10, it will be stored in refrigerator at the operative clinic to avoid exposure to high temperature or sunlight.
  Interventions: Combination Product: fluoride varnish (Bifluorid 10)

INTERVENTIONS:
Combination Product: Sylc — a dry powder (calcium sodium phosphosilicate), based on NovaMin powder. Bottle of small and coarse particles will be used for the treatment
  Other Names: Sylc bioactive glass
  Arms: sylc bioactive glass
Combination Product: fluoride varnish (Bifluorid 10) — It is a rapid- drying suspension of equal amounts of sodium fluoride and calcium fluoride.
  Other Names: Bifluorid 10
  Arms: fluoride varnish (Bifluorid 10)

SUMMARY:
Will the use of Bioactive glass with air abrasion technology (Sylc) compared to Fluoride Varnish (Biflourid 10) affects the degree of pain in patients complaining from hypersensitivity due to non-carious lesions?

DETAILED DESCRIPTION:
* Population: Patients complaining from Dentin Hypersensitivity due to non-carious lesions.
* Intervention: Sylc, Air Abrasion Bioactive glass (Denfotex Research Ltd.)
* Comparison: BiFlourid 10, Fluoride Varnish (VOCO, Germany)
* Outcome measures: Dentin Hypersensitivity

Outcome name Measuring device Measuring unit Dentin Hypersensitivity

* Thermal
* Tactile
* Evaporative

ELIGIBILITY:
Inclusion Criteria:

* Males or females.
* Age: 18-70 years old.
* Patients with good oral hygiene.
* Co-operative patients who show interest to participate in the study.

Exclusion Criteria:

* Patients with bad oral hygiene.
* Patients with orthodontic appliances, or bridge work that might interfere with evaluation.
* Patients who did any periodontal surgeries within the previous 6 months.
* Patients who are allergic to any ingredients will be used in the study.
* Pregnant and lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Pain due to dentin hypersensitivity (evaporative stimulus) | 2 minutes after treatment
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by air blast measured by a 10 cm visual analogue scale VAS

SECONDARY OUTCOMES:
Pain due to dentin hypersensitivity (evaporative stimulus) | 1 week
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by air blast measured by a 10 cm visual analogue scale VAS
Pain due to dentin hypersensitivity (evaporative stimulus) | 2 weeks
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by air blast measured by a 10 cm visual analogue scale VAS
Pain due to dentin hypersensitivity (evaporative stimulus) | 3 weeks
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by air blast measured by a 10 cm visual analogue scale VAS
Pain due to dentin hypersensitivity (evaporative stimulus) | 4 weeks
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by air blast measured by a 10 cm visual analogue scale VAS
Pain due to dentin hypersensitivity (evaporative stimulus) | 6 months
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by air blast measured by a 10 cm visual analogue scale VAS
Pain due to dentin hypersensitivity (evaporative stimulus) | 12 months
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by air blast measured by a 10 cm visual analogue scale VAS
Pain due to dentin hypersensitivity (tactile stimulus) | 2 minutes after treatment
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by tactile stimulation with a probe measured by a 10 cm visual analogue scale VAS
Pain due to dentin hypersensitivity (tactile stimulus) | 1 week
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by tactile stimulation with a probe measured by a 10 cm visual analogue scale VAS
Pain due to dentin hypersensitivity (tactile stimulus) | 2 weeks
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by tactile stimulation with a probe measured by a 10 cm visual analogue scale VAS
Pain due to dentin hypersensitivity (tactile stimulus) | 3 weeks
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by tactile stimulation with a probe measured by a 10 cm visual analogue scale VAS
Pain due to dentin hypersensitivity (tactile stimulus) | 4 weeks
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by tactile stimulation with a probe measured by a 10 cm visual analogue scale VAS
Pain due to dentin hypersensitivity (tactile stimulus) | 6 months
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by tactile stimulation with a probe measured by a 10 cm visual analogue scale VAS
Pain due to dentin hypersensitivity (tactile stimulus) | 12 months
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by tactile stimulation with a probe measured by a 10 cm visual analogue scale VAS
Pain due to dentin hypersensitivity (thermal stimulus) | 2 minutes after treatment
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by cold water measured by a 10 cm visual analogue scale VAS
Pain due to dentin hypersensitivity (thermal stimulus) | 1 week
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by cold water measured by a 10 cm visual analogue scale VAS
Pain due to dentin hypersensitivity (thermal stimulus) | 2 weeks
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by cold water measured by a 10 cm visual analogue scale VAS
Pain due to dentin hypersensitivity (thermal stimulus) | 3 weeks
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by cold water measured by a 10 cm visual analogue scale VAS
Pain due to dentin hypersensitivity (thermal stimulus) | 4 weeks
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by cold water measured by a 10 cm visual analogue scale VAS
Pain due to dentin hypersensitivity (thermal stimulus) | 6 months
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by cold water measured by a 10 cm visual analogue scale VAS
Pain due to dentin hypersensitivity (thermal stimulus) | 12 months
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by cold water measured by a 10 cm visual analogue scale VAS

CONTACTS AND LOCATIONS:
Overall Officials: Dina E Mohamed, Master, Principal Investigator — Assistant lecturer, Conservative Dentistry Department, Faculty of Dentistry, Cairo University
Locations (1):
- Faculty of dentistry, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided